CLINICAL TRIAL: NCT00764803
Title: Post-Market Study: The Efficacy of the 3DKnee™ System vs. the MJS Knee System
Brief Title: 3DKnee™ System vs. the MJS Knee System
Status: Terminated | Type: Observational
Why Stopped: Corporate decision to discontinue distribution of MJS Knee.
Sponsor: Encore Medical, L.P. (Industry)
Responsible Party: Jane M. Jacob Ph.D., DJO Surgical
Other Study IDs: PS - 702
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2010-03-11 (Estimated); Status verified 2010-03

CONDITIONS: Rheumatoid Arthritis; Traumatic Arthritis; Joint Disease Secondary to Osteoarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 2: Subjects who meet the indications for use and are implanted with the Encore MJS™ Knee System.
  Interventions: Device: Encore MJS™ Knee System
- 1: Subjects who meet the indications for and are implanted with the Encore 3DKnee™ system.
  Interventions: Device: Encore 3DKnee™ system

INTERVENTIONS:
Device: Encore 3DKnee™ system — Subjects with rheumatoid arthritis, traumatic arthritis or osteoarthritis who were implanted with the Encore 3DKnee™ system and willing to participate in the study.
  Groups: 1
Device: Encore MJS™ Knee System — Subjects with rheumatoid arthritis, traumatic arthritis or osteoarthritis who were implanted with the Encore MJS™ Knee system and willing to participate in the study.
  Groups: 2

SUMMARY:
The purpose of this study is to compare the survivorship and efficacy of the Encore 3DKnee™ system with that of the Encore MJS™ Knee System in a group of 600 patients for whom data collection is already under way.

DETAILED DESCRIPTION:
The purpose of this study is to compare the survivorship and efficacy of the Encore 3DKnee™ system with that of the Encore MJS™ Knee System in a group of 600 patients for whom data collection is already under way. Approximately 300 patients have already received the MJS™ knee system and data, as described below, has been collected for these patients over a period of two years. A second group of 300 patients will receive the Encore 3DKnee™ system over the next two years, and equivalent data will be collected for these individuals. A portion of the data has been collected over the past year, and now we would like to obtain permission from the patients to analyze these data as well as collect an additional year of data.

ELIGIBILITY:
Inclusion Criteria:

* This must be a primary knee replacement on this knee.
* Patient is over 18 years of age or older
* Patients must have one of the following

  * rheumatoid or traumatic arthritis OR
  * joint disease secondary to osteoarthritis
* Patient is likely to be available for evaluation for the duration of the study
* Able and willing to sign the informed consent and follow study procedures
* Patient is not pregnant

Exclusion Criteria:

* Is younger than 18 years of age
* If there has been a total knee replacement on this knee in the past (no revisions allowed in study)
* Overt infection
* Alcoholism or other addictions
* Muscular, neurological or vascular deficiencies which compromise the affected extremity
* Obesity
* Marked bone loss
* Materials sensitivity
* Prisoner
* Mental conditions that may interfere with the patient's ability to give an informed consent or willingness to fulfill the study requirements
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who meet either the indications for use of the 3DKnee or the MJS knee system. Subjects must also meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The survivorship and efficacy of the Encore 3DKnee™ system with that of the Encore MJS™ Knee System | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: D. Kevin Lester, M.D., Principal Investigator — Center for Excellence
Locations (1):
- Center for Excellence, Fresno, California, United States

REFERENCES:
- See also: Sponsor company home page — http://www.djosurgical.com